CLINICAL TRIAL: NCT04266639
Title: Rheo-Erythrocrine Dysfunction as a Biomarker for RIC Treatment in Acute Ischemic Stroke - Pilot, Single-center, Randomized, Patient-assessor Blinded, Sham-controlled Study
Brief Title: Rheo-Erythrocrine Dysfunction as a Biomarker for RIC Treatment in Acute Ischemic Stroke
Acronym: ENOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grethe Andersen (Other)
Responsible Party: Sponsor-Investigator, Grethe Andersen, Professor, DMSc, Senior Consultant, MD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENOS
Record Dates: First submitted 2020-02-03; First posted 2020-02-12 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Stroke, Acute; Ischemic Stroke; Cerebrovascular Disorders; Central Nervous System Diseases
Keywords: Remote Ischemic Conditioning; Neuroprotection
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Pilot, Single-center, Randomized, Patient-assessor blinded, Sham-controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote Ischemic Conditioning (Active Comparator): Remote Ischemic Conditioning (RIC) is applied during the in-hospital phase using an automated RIC device.
  Treatment characteristics: Five cycles (50 minutes), each consisting of five minutes of cuff inflation followed by five minutes of cuff deflation. The cuff pressure will be 200 mmHg; if initial systolic blood pressure is above 175 mmHg, the cuff is automatically inflated to 35 mmHg above the systolic blood pressure.
  * Initial Remote Ischemic Conditioning: < 2 hours from inclusion
  * Remote Ischemic Postconditioning: twice daily for 7 days
  Usual care with or without acute reperfusion therapy
  Interventions: Device: Remote Ischemic Conditioning
- Sham - Remote Ischemic Conditioning (Sham Comparator): Sham Remote Ischemic Conditioning (Sham-RIC) is applied during the in-hospital phase using an automated Sham-RIC device.
  Treatment characteristics: Five cycles (50 minutes), each consisting of five minutes of cuff inflation followed by five minutes of cuff deflation. The cuff pressure will be always be 20 mmHg.
  * Initial Sham Remote Ischemic Conditioning: < 2 hours from inclusion
  * Sham Remote ischemic Postconditioning: twice daily for 7 days
  Usual care with or without acute reperfusion therapy.
  Interventions: Device: Sham Remote Ischemic Conditioning
- Controls (No Intervention): The control group will not receive treatment with Remote Ischemic Conditioning.

INTERVENTIONS:
Device: Remote Ischemic Conditioning — RIC is commonly achieved by inflation of a blood pressure cuff to induce 5-minute cycles of limb ischemia alternating with 5 minutes of reperfusion
  Arms: Remote Ischemic Conditioning
Device: Sham Remote Ischemic Conditioning — Sham Comparator (Sham-RIC)
  Arms: Sham - Remote Ischemic Conditioning

SUMMARY:
This study aims to investigate whether Remote Ischemic Conditioning (RIC) improves rheo-erythrocrine dysfunction in acute ischemic stroke

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability worldwide. Of all strokes, 85% are ischemic strokes caused by a thrombus or an embolus. The additional 15% are caused by hemorrhage. Currently the only approved treatments for ischemic strokes are thrombolysis given within 4.5 hours and thrombectomy performed within 6 hours of symptom onset - in some cases up to 24 hours. The majority of stroke patients are not however eligible for acute reperfusion therapy, mainly due to time constrains and late presentation. Novel neuroprotective strategies available for all stroke patients are thus urgently needed.

Remote Ischemic Conditioning (RIC) is a simple intervention in which transient ischemia is induced in an extremity by repetitive inflation-deflation of a blood pressure cuff. It remains uncertain exactly how the protective effect of RIC is transmitted and communicated between the extremity and the brain. Both humoral, immunological and neuronal pathways seem to be involved. Treatment with RIC and has proven to be a safe, feasible and low-cost treatment in clinical settings.

Biomarkers of the RIC treatment is a new area of stroke research and are important to establish in order to assess and predict responders of the conditioning treatment. Rheo-erythrocrine dysfunction of the Red Blood Cell (RBC) is a novel biomarker in both ischemic strokes in general and on the effect of RIC. Red Blood Cells with a diameter of 6-8 μm must be highly deformable in order to deliver oxygen to brain tissue by travelling through micro vessels with a diameter of just 2-3 μm. RBC's can carry nitric oxide as NO2-/s-nitrosylated proteins. These proteins improve RBC deformability and induce hypoxic vasodilation thereby improving passage through the microvasculature. RBC's also express Erythrocyte Nitric Oxide Synthase 3, which regulate the rheo-erythrocrine function. Erythrocyte Nitric Oxide Synthase 3 is activated by shear stress and provide an extra source of NO for hypoxic vasodilation. Preliminary data have shown that experimental stroke on mice seems to cause a rheo-erythrocrine dysfunction of the RBC's leading to a loss of deformability. The RBC's become rigid, which can lead to occlusion of micro vessels in the brain and further ischemic damage. Loss of deformability can be measured as a reduced Elongation Index (EI) by ektacytometry and may be attenuated by RIC.

ELIGIBILITY:
STROKE PATIENTS

Inclusion Criteria:

* Onset to randomization < 48 hours
* Independent in daily living (mRS 0-2)
* Legal competent
* Ambulatory
* Documented ischemic stroke on baseline MRI

Exclusion Criteria:

* Prior stroke, dementia or other known neurological condition Pregnancy
* Contraindications to MRI
* Investigators discretion
* Known upper extremity peripheral arterial stenosis Diabetes

CONTROLS

Inclusion Criteria:

* Independent in daily living (mRS 0-2) Ambulatory
* Legal competent
* Non vascular diagnosis (e.g. epilepsy, migraine etc.)

Exclusion Criteria

* Prior stroke, dementia or other known neurological condition
* Pregnancy
* Contraindications to MRI
* Investigators discretion
* Known upper extremity peripheral arterial stenosis Diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
RBC deformability will serve as a biomarker of the conditioning response and predictor of the clinical outcome in stroke patients. | 1 week
  RBC deformability is measured as Deformability or Elongation Index (DI or EI, Rheoscan AnD-300, RheoMeditech, South Chorea). A higher EI at the optimum viscosity (300 Osmolality) indicates highly deformable RBCs indicative of better microcirculation, while a lower EI indicates rigid RBC's. Briefly, 6 µL of heparinized or EDTA treated fresh blood is mixed with 600-µL of polyvinylpyrrolidone (PVP) solution (300 Osm) and transferred to a disposable kit. The kit is placed inside the laser-assisted ectacytometer for automated read out, data and image collection as per the vendor's instructions.
RBC deformability will serve as a biomarker of the conditioning response and predictor of the clinical outcome in stroke patients | 1 week
  For measurement of shear stress, 0,5 mL of heparinized or EDTA treated fresh blood is mixed with 600-µL of polyvinylpyrrolidone (PVP) solution (300 Osm) and transferred to a disposable kit. The kit is placed inside the laser-assisted ectacytometer for automated read out, data and image collection as per the vendor's instructions.

SECONDARY OUTCOMES:
Nitric oxide quantification using DAF-FM-Diacetate flowcytometry as a biomarker of the conditioning response | 1 week
  Analytical flowcytometry with DAF-FM-Diacetate (4-Amino-5-Methylamino-2',7'-Difluorofluorescein Diacetate) on wholeblood samples
Nitric oxide quantification using DAF-FM-Diacetate flowcytometry as a predictor of the short term clinical outcome in stroke patients | 1 week
  Analytical flowcytometry with DAF-FM-Diacetate (4-Amino-5-Methylamino-2',7'-Difluorofluorescein Diacetate) on wholeblood samples
RBC deformability presentation across stroke subtypes | 1 week
  Ektacytometry (see primary outcome)
RBC deformability in relation to infarct size/stroke severity | 1 week
  Ektacytometry (see primary outcome)
RBC erythrocrine dysfunction (NOS3) presentation across stroke subtypes | 9 months
  Comparison of RBC Nitric Oxide Synthestase 3 activation (flowcytometry) across stroke subtypes.
RBC erythrocrine dysfunction (nitric oxide) presentation across stroke subtypes | 9 months
  Comparison of nitric oxide estimation (chemiluminescence) across stroke subtypes
RBC erythrocrine dysfunction (NOS3) in relation to infarct size/stroke severity | 9 months
  Level of RBC Nitric Oxide Synthestase 3 activation (flowcytometry)
RBC erythrocrine dysfunction (nitric) in relation to infarct size/stroke severity | 9 months
  Level of nitric oxide estimation (chemiluminescence)
Difference in 7 days cognitive impairment between treatment groups | 1 week
  Difference between baseline Montreal Cognitive Assessment (MoCA) score and day 7 MoCA score.
  MoCA is a 1-page (healthcare administered), 0-30-point test (30 is the best score), administrable in ≈10 minutes. The test evaluates different domains: visuospatial abilities, executive functions, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space.
RBC erythrocrine dysfunction and deformability as a marker for difference in 7 days cognitive impairment (MoCA scale) | 9 months
  Cognitive impairment is measured using the Montreal Cognitive Assessment scale (MoCA), which is a 1-page (healthcare administered), 0-30-point test (30 is the best score), administrable in ≈10 minutes. The test evaluates different domains: visuospatial abilities, executive functions, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space
Circulating microRNA profile of RIC-induced neuroprotection | 9 months
  MicroRNAs will be identified with Illumina next-generation sequencing using the TruSeq Small RNA Sample Preparation kit. The output will be miRNA expression levels for each sample, which will form the basis for a miRNA differential analysis where miRNAs with statistically significant expression changes will be found
Extracellular vesicle profile of RIC-induced neuroprotection | 9 months
  Extracellular vesicles (EVs, also known as exosomes) will be isolated from plasma samples before characterization of surface markers and content. Protein characterization will be done using ELISA and Western blots in addition to array techniques. To broaden the feasibility of finding stroke type specific EV surface markers, we will utilize recombinant antibody library techniques to find novel disease binders with the potential of diagnosing stroke types in blood samples. Nucleic acid (DNA and RNA including miRNA) content of EVs will be analyzed using next generation sequencing (NGS) and qRT-PCR
Circulating microRNA as a marker for difference in 7 days cognitive impairment (MoCA score) | 9 months
  Cognitive impairment is measured using the Montreal Cognitive Assessment scale (MoCA), which is a 1-page (healthcare administered), 0-30-point test (30 is the best score), administrable in ≈10 minutes. The test evaluates different domains: visuospatial abilities, executive functions, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space
Extracellular vesicle profile as a marker for RBC erythrocrine dysfunction and deformability | 9 months
  Extracellular vesicles (EVs, also known as exosomes) will be isolated from plasma samples before characterization of surface markers and content. To broaden the feasibility of finding stroke type specific EV surface markers, we will utilize recombinant antibody library techniques to find novel disease binders with the potential of diagnosing stroke types in blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Andersen, MD, DMSc, Principal Investigator — Aarhus University Hospital, Department of Neurology
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT04266639/Prot_000.pdf